CLINICAL TRIAL: NCT06619678
Title: An Open-Label Study to Assess the Two-Way Interaction Between Multiple Weekly Doses of MK-8507 and Single Doses of Islatravir (MK-8591) in Healthy Adult Participants
Brief Title: A Study of MK-8507 and Islatravir (MK-8591) in Healthy Adult Participants (MK-8507-016)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8507-016; MK-8507-016 (Other: MSD)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — ulonivirine; islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Islatravir+MK-8507 (Experimental): Period 1: Participants receive single dose of Islatravir on Day 1. Period 2: Participants receive single dose of MK-8507 on Days 1 and Days 8. Period 3: Participants receive single dose of Islatravir and single dose of MK-8507 on Day 1, 7 days after the Day 8 dose of MK-8507, during Period 2. Participants will receive additional MK-8507 single doses on Days 8, 15, 22, and 29.
  Interventions: Drug: MK-8507; Drug: Islatravir

INTERVENTIONS:
Drug: MK-8507 — Oral administration
Drug: Islatravir — Oral administration
  Other Names: ISL; MK-8591

SUMMARY:
The main goals of this study are to learn what happens to Islatravir or MK-8507 in a person's body over time. Researchers will compare Islatravir given alone to Islatravir given with MK-8507. Researchers will also compare MK-8507 given alone to MK-8507 given with Islatravir.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer with protocol specified exceptions

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Islatravir Metabolite | At designated timepoints (up to approximately 43 days)
  Blood samples will be collected to determine the AUC0-Inf of Islatravir metabolite.
Area Under the Concentration-Time Curve from Time 0 to 168 hours (AUC0-168hrs) of Islatravir Metabolite | At designated timepoints (up to approximately 168 hours)
  Blood samples will be collected to determine the AUC0-168hrs of Islatravir metabolite.
Maximum Concentration (Cmax) of Islatravir Metabolite | At designated timepoints (up to approximately 43 days)
  Blood samples will be collected to determine Cmax of Islatravir metabolite.
Plasma Concentration at 168 Hours (C168) of Islatravir Metabolite | At designated timepoints (up to approximately 168 hours)
  Blood samples will be collected to determine the C168 of Islatravir metabolite.
Time to Maximum Concentration (Tmax) of Islatravir Metabolite | At designated timepoints (up to approximately 43 days)
  Blood samples will be collected to determine the Tmax of Islatravir metabolite.
Apparent Terminal Half-life (t1/2) of Islatravir Metabolite | At designated timepoints (up to approximately 43 days)
  Blood samples will be collected to determine the t1/2 of Islatravir metabolite.
AUC0-Inf of Islatravir | At designated timepoints (up to approximately 22 days)
  Blood samples will be collected to determine the AUC0-Inf of Islatravir.
AUC0-168hrs of Islatravir | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the AUC0-168hrs of Islatravir.
Cmax of Islatravir | At designated timepoints (up to approximately 22 days)
  Blood samples will be collected to determine Cmax of Islatravir.
C168 of Islatravir | At designated timepoints (up to approximately 168 hours)
  Blood samples will be collected to determine the C168 of Islatravir.
Tmax of Islatravir | At designated timepoints (up to approximately 22 days)
  Blood samples will be collected to determine the Tmax of Islatravir.
t1/2 of Islatravir | At designated timepoints (up to approximately 22 days)
  Blood samples will be collected to determine the t1/2 of Islatravir.
Apparent clearance (CL/F) of Islatravir | At designated timepoints (up to approximately 22 days)
  Blood samples will be collected to determine the CL/F of Islatravir.
Apparent Volume of Distribution During Terminal Phase (Vd/F) of Islatravir | At designated timepoints (up to approximately 22 days)
  Blood samples will be collected to determine the Vd/F of Islatravir.
AUC0-168hrs of MK-8507 | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the AUC0-168hrs of MK-8507.
Cmax of MK-8507 | At designated timepoints (up to approximately 15 days)
  Blood samples will be collected to determine Cmax of MK-8507.
C168 of MK-8507 | At designated timepoints (up to approximately 168 hours)
  Blood samples will be collected to determine the C168 of MK-8507.
Tmax of MK-8507 | At designated timepoints (up to approximately 15 days)
  Blood samples will be collected to determine the Tmax of MK-8507.
t1/2 of MK-8507 | At designated timepoints (up to approximately 15 days)
  Blood samples will be collected to determine the t1/2 of MK-8507.
CL/F of MK-8507 | At designated timepoints (up to approximately 15 days)
  Blood samples will be collected to determine the CL/F of MK-8507.
Vd/F of MK-8507 | At designated timepoints (up to approximately 15 days)
  Blood samples will be collected to determine the Vd/F of MK-8507.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 5 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 5 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com